CLINICAL TRIAL: NCT00872352
Title: Phase 3 Study to Evaluate Bortezomib Induced Peripheral Neuropathy of Multiple Myeloma (MM) Patients.
Brief Title: Evaluation of Bortezomib Induced Peripheral Neuropathy of Multiple Myeloma (MM) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: HusamGhoti, MD, Hematology Dept., Wolfson MC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 1.1
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma; Peripheral Neuropathy
Keywords: Multiple Myeloma; Bortezomib; Peripheral Neuropathy; evaluation; evaluation of electrophysiological changes related to the dose and time of bortezomib administration; investigation of correlation between the incidence of BIPN and the subtype of myeloma
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: EMG — Nerve conduction study will be consisted of sequential evaluation of the motor nerves: median, ulnar, peroneal and tibial; and the sensory nerves: median, ulnar, superficial peroneal and sural nerves using a standardized protocol

SUMMARY:
In the present study we are planning to study electrophysiological changes related to the dose and time of bortezomib administration in newly diagnosed patients with MM, during the first months of treatment and 6 months after ending. In addition a possible correlation between the incidence of BIPN and the subtype of myeloma and other risk factors will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18
* Patients with Multiple Myeloma stage II, III (Durie and Salmon staging) prior to Bortezomib Therapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Be willing and able to comply with the protocol treatment for the duration of the study
* Patient's written informed consent

Exclusion Criteria:

* Multiple Myeloma on progression
* Incidence of Relapsed or Refractory Myeloma
* Patients with the existing neuropathy at the time of the diagnosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
A dose-related neurotoxic effect of bortezomib will be determined through regression analysis with the change in TNSr as the dependent variable Bortezomib doses will use as independent variables. | 3 months

SECONDARY OUTCOMES:
To accommodate the dose of bortezomib with the progression of Peripheral Neuropathy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Rachmilewitz, MD, Study Director — Head of Hematology, Wolfson MC, Holon, Israel
Locations (1):
- Wolfson MC, Holon, Holon, Israel